CLINICAL TRIAL: NCT01418157
Title: Double Blind, Placebo Controlled Randomised Trial of Acetazolamide Versus Placebo in the Prevention of Acute Mountain Sickness During Rapid Ascent
Brief Title: A Trial of Acetazolamide Versus Placebo in Preventing Mountain Sickness During Rapid Ascent
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Oxford University Clinical Research Unit, Vietnam (Other)
Collaborators: University of Oxford (Other); Wellcome Trust (Other); Mountain Medicine Society of Nepal (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 04NP
Record Dates: First submitted 2011-08-08; First posted 2011-08-16 (Estimated); Last update posted 2013-06-24 (Estimated); Status verified 2013-06

CONDITIONS: Acute Mountain Sickness
Keywords: Acute mountain sickness; Rapid ascent; High altitude headache; Mountain Medicine Society Nepal
MeSH Terms: conditions — Altitude Sickness | interventions — Acetazolamide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Acetazolamide (Active Comparator)
  Interventions: Drug: Acetazolamide
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Acetazolamide — 125 mg twice daily until 4380 meters altitude
  Arms: Acetazolamide
Drug: Placebo — Twice daily
  Arms: Placebo

SUMMARY:
Acute mountain sickness is a common ailment in people venturing over 2500 m altitude. Pilgrims to high altitudes are at an added risk since they are unaware and they gain height faster than the recommendations. Acetazolamide is the standard treatment and prophylaxis of acute mountain sickness. There are no randomized controlled trials that have studied protective effects of Acetazolamide in rapid ascent, and there are few conflicting studies regarding this matter.

This study is a randomized, double blinded, placebo controlled trial of Acetazolamide versus placebo in 380 healthy individuals travelling to Gosaikunda Lake of Nepal in rates of ascent that are faster than the recommendations. Acetazolamide 125 mg twice daily and a placebo will be randomly assigned for 3 days and participants will be assessed at 3 stations.

This study will undertake to establish the role of Acetazolamide in Rapid Ascent and will be the first RCT done in this issue.

The investigators hypothesize that Acetazolamide 125mg twice daily given before rapid ascent to high altitude in Nepalese pilgrims will not be superior to placebo in decreasing both the incidence and severity of acute mountain sickness.

ELIGIBILITY:
Inclusion Criteria:

* Nepalese national
* Aged 18 to 65
* Travelling directly from Dhunche to Gosainkunda
* Rapid ascent as defined by ascent within 3 days

Exclusion Criteria:

* Use of any drugs for the prevention of altitude sickness or headache
* Current illness
* Current altitude sickness (more than one mild symptom on the Lake Louise Questionnaire (LLQ), or oxygen saturation less than 75%
* Known to be pregnant or cannot exclude the possibility of being pregnant, or have missed menses by over 7 days
* One night within the last 30 days spent at an altitude of 4500 metres or above
* Residents of altitude more than 2500m
* A known drug allergy to sulfonamides.
* Treatment with any of the following in the last 2 days: acetazolamide (Diamox®), steroids (dexamethasone/decadron, prednisone), theophylline or diuretics (Lasix®), ibuprofen/motrin, naprosyn/naproxen, aspirin or acetaminophen.
* Any serious intracranial abnormalities such as history of brain tumours or pseudotumour cerebri
* Known severe uncontrolled headache syndrome
* Diagnosed renal function impairment, diabetes, cirrhosis of liver or liver dysfunction

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 380 (Actual)
Dates: Start 2011-08; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Diagnosis of acute mountain sickness | Upon reaching an altitude of 3300m, average expected time is 1 day
  A diagnosis of AMS requires a score of three or greater on the Lake Louise Acute Mountain Sickness Questionnaire with the mandatory presence of headache and at least one of the following symptoms: dizziness or light-headedness, fatigue, gastrointestinal (GI) symptoms (nausea/vomiting), or difficulty sleeping.
Diagnosis of acute mountain sickness | Upon reaching an altitude of 4380m, average expected time is 3 days
  A diagnosis of AMS requires a score of three or greater on the Lake Louise Acute Mountain Sickness Questionnaire with the mandatory presence of headache and at least one of the following symptoms: dizziness or light-headedness, fatigue, gastrointestinal (GI) symptoms (nausea/vomiting), or difficulty sleeping.

SECONDARY OUTCOMES:
Blood oxygen saturation | Upon reaching an altitude of 3300m, average expected time is 1 day
  Percent
Heart rate | Upon reaching an altitude of 3300m, average expected time is 1 day
  Beats per minute
High altitude headache | Upon reaching an altitude of 3300m, average expected time is 1 day
  High altitude headache severity will be scored in milimeters based on patient markings on a visual analog scale. The headache score will be identified on the designated Lake Louise Questionnaire.
Blood oxygen saturation | Upon reaching an altitude of 4380m, average expected time is 3 days
  Percent
Heart rate | Upon reaching an altitude of 4380m, average expected time is 3 days
  Beats per minute
High altitude headache | Upon reaching an altitude of 4380m, average expected time is 3 days
  High altitude headache severity will be scored in millimeters based on patient markings on a visual analog scale. The headache score will be identified on the designated Lake Louise Questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Buddha Basnyat, MD PhD, Principal Investigator — University of Oxford
Locations (1):
- Oxford University Clinical Research Unit Nepal, Kathmandu, Nepal

REFERENCES:
- [Result] Gertsch JH, Corbett B, Holck PS, Mulcahy A, Watts M, Stillwagon NT, Casto AM, Abramson CH, Vaughan CP, Macguire C, Farzan NN, Vo BN, Norvelle RJ, May K, Holly JE, Irons H, Stutz AM, Chapagain P, Yadav S, Pun M, Farrar J, Basnyat B. Altitude Sickness in Climbers and Efficacy of NSAIDs Trial (ASCENT): randomized, controlled trial of ibuprofen versus placebo for prevention of altitude illness. Wilderness Environ Med. 2012 Dec;23(4):307-15. doi: 10.1016/j.wem.2012.08.001. Epub 2012 Oct 24. PMID 23098412
- See also: Mountain Medicine Society Nepal — http://mmsn.org.np/
- See also: Oxford University Clinical Research Unit Viet Nam — http://www.oucru.org
- See also: Oxford University Clinical Research Unit Nepal — http://www.tropicalmedicine.ox.ac.uk/nepal
- See also: Trial Informed Consent Form, approvals and additional information — http://www.oucru.org/index.php?option=com_content&view=article&id=336&Itemid=111&lang=en